CLINICAL TRIAL: NCT04697251
Title: Application of Forced Oscillation Technique in Infancy
Brief Title: Infant Forced Oscillations Technique (iFOT)
Acronym: iFOT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Patras (Other)
Responsible Party: Principal Investigator, Fouzas Sotirios, Assistant Professor of Pediatrics, University of Patras
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 28292/20201103
Record Dates: First submitted 2021-01-02; First posted 2021-01-06 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Respiratory Function Tests; Respiratory Disease; Infant, Newborn, Disease
MeSH Terms: conditions — Respiration Disorders; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FOT measurements (Other): FOT measurements in newborns and small infants
  Interventions: Diagnostic Test: FOT measurements in newborns and small infants

INTERVENTIONS:
Diagnostic Test: FOT measurements in newborns and small infants — Measurements will be performed using the device TremoFlo N-100, at bedside, with the infant in the supine position during quiet natural sleep. After proper cleaning and decontamination, the face mask of the device will be preheated at 37oC (to avoid awakening) and will be placed on infant's face. The duration of each measurement will be predetermined at 10 s. At least 3 technically acceptable measurements will be performed per infant, with 30 s intervals between them. The validity of each measurement will be assessed according to the coherence function (automatically determined by the operating system of the device).

SUMMARY:
The aim of this study is the implementation of Forced Oscillations Technique (FOT) in newborns and small infants using a novel commercially available device.

The objective is to assess the feasibility of the method, provide normative data for the first months of life and describe short- and long-term changes in neonatal respiratory disorders.

The study population will consist of term and preterm newborns admitted to the Neonatal Intensive Care Unit (NICU) or the Well-Baby Nursery of the University Hospital of Patras, Greece. It is estimated that 200 full-term and 150 preterm newborns will be enrolled during a period of 36 months (March 2021 - September 2022).

Measurements will be performed using the TremoFlo N-100 via a face mask, with the infant in the supine position during natural sleep. At least 3 technically acceptable measurements (duration 10s each) will be obtained, as follows:

* Healthy full-term neonates: postnatal days 1, 2, 3 and at discharge
* Preterm neonates: NICU admission, postnatal days 1, 2 and 3, and on the first day of each additional gestational week until discharge

All participants will be also measured at the age of 3, 6 and 12 months.

DETAILED DESCRIPTION:
INTRODUCTION Pulmonary function testing during early infancy requires sophisticated equipment, specialized personnel and proper patient's preparation. As a result, lung function testing in newborns and small infants is limited to few highly specialized centers.

The forced oscillations technique (FOT) uses complex pressure signals generated by an external device at the airway opening. The pressure waves are transmitted through the airway tree during tidal breathing and force the anatomical structures of the respiratory system to oscillate. From subsequent pressure and flow signal analysis, the total resistance (Rrs) and reactance (Xrs) of the respiratory system are calculated. The latter relates mainly to the elastic properties of the lung parenchyma and the inertia of the column of air in the airways. Both Rrs and Xrs depend on the frequency of oscillation; lower frequencies (range 5-10Hz) provide information on the mechanical properties of smaller airways and vice versa. FOT measurements can be performed fast (usually in less than 30 s), at the bedside, and do not require patient's cooperation. Therefore, FOT is being viewed as an attractive and promising pulmonary function technique for young infants and newborns.

To date, the introduction of infant FOT in routine clinical practice has been limited due to lack of suitable devices and normative data. Studies based on in-build FOT equipment have shown that the application of the method in small infants is feasible. A recent study, in which a modified commercially available device (Tremoflo C-100, THORASYS Thoracic Medical Systems Inc. Montreal, Canada) was used, also supports the feasibility of the method.

OBJECTIVE The aim of this study is the implementation of FOT in newborns and small infants using a novel commercially available device (Tremoflo N-100, THORASYS), specifically released for this age range.

Our objectives are: a) to assess the feasibility of the method and the repeatability of FOT measurements in newborns and small infants, b) to provide normative data for the first months of life in relation to various parameters (e.g. gender, age, somatometrics, etc) and, c) to describe short- and long-term and Rrs and Xrs changes in neonatal respiratory disease (e.g. respiratory distress syndrome, bronchopulmonary dysplasia, etc).

METHODS Population The study population will consist of term and preterm newborns admitted to the Neonatal Intensive Care Unit (NICU) or the Well-Baby Nursery of the University Hospital of Patras, Greece. It is estimated that 200 full-term and 150 preterm newborns will be enrolled during a period of 36 months (March 2021 - September 2022).

The parents of all infants will provide written informed consent prior to enrollment. The study has been approved by the Research and Ethics Committee of the hospital (decision no. 451/12.11.2020).

Measurements Measurements will be performed using the TremoFlo N-100, at bedside, with the infant in the supine position during quiet natural sleep. The device will be calibrated daily, according to manufacturer's instructions. After proper cleaning and decontamination, the face mask of the device will be preheated at 37oC (to avoid awakening) and will be placed on infant's face. The duration of each measurement will be predetermined at 10 s. At least 3 technically acceptable measurements will be performed per infant, with 30 s intervals between them. The validity of each measurement will be assessed according to the coherence function (automatically determined by the operating system of the device).

Protocol

FOT measurements will be scheduled according to the target population, as follows:

* In healthy full-term neonates, measurements will be obtained on postnatal days 1, 2, 3 and at discharge. Parents will be asked and scheduled to repeat testing at the age of 3, 6 and 12 months.
* In preterm neonates without respiratory disease, measurements will be performed on NICU admission, on postnatal days 1, 2 and 3, and on the first day of each additional gestational week until discharge. For example, a preterm neonate with gestational age 331/7, will be measured at 331/7, 332/7, 333/7, 334/7, 34, 35, 36, etc. Parents of preterm newborns will be also asked and scheduled to repeat testing at the age of 3, 6 and 12 months.
* In preterm neonates with respiratory distress syndrome (RDS) the measurements will be obtained on NICU admission and at 6 and 12 hours after surfactant administration. Thereafter, the same protocol with preterm neonates without respiratory disease will be applied. In mechanically ventilated infants the measurements will be performed via the endotracheal tube, but only if their clinical condition permits FOT testing. In such cases, the device will be calibrated in advance using an endotracheal tube of the same internal diameter, material and length as that positioned on the neonate.

EXPECTED RESULTS AND BENEFITS The study is expected to confirm the feasibility of FOT in newborns and small infants (in NICU or outpatient settings) and, most important, to reveal a series of technical/practical details that may improve the applicability of the method in clinical practice. Finally, the study will provide normative data for this age range, and will assess Rrs and Xrs changes in various respiratory disorders of the neonatal period and early infancy.

ELIGIBILITY:
Inclusion Criteria:

* Newborns cared for in the NICU and well-baby nursery of the University Hospital of Patras, Greece.
* Parental written informed consent.

Exclusion Criteria:

* Major respiratory, cardiovascular or other condition that does not permit FOT measurements at the predetermined time points.
* Any infectious disorder with increased risk of contamination.
* Orofacial anomalies (e.g. genetic syndromes) that do not permit proper application of the face mask.

Ages: 1 Day to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 350 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Respiratory resistance (Rrs) - Term newborns | Postnatal day 1.
  Rrs at multiple frequencies (FOT) in term infants
Respiratory resistance (Rrs) - Term newborns | Postnatal day 2.
  Rrs at multiple frequencies (FOT) in term infants
Respiratory resistance (Rrs) - Term newborns | Postnatal day 3.
  Rrs at multiple frequencies (FOT) in term infants
Respiratory resistance (Rrs) - Term newborns | On the day of discharge.
  Rrs at multiple frequencies (FOT) in term infants
Respiratory reactance (Xrs) - Term newborns | Postnatal day 1.
  Xrs at multiple frequencies (FOT) in term infants
Respiratory reactance (Xrs) - Term newborns | Postnatal day 2.
  Xrs at multiple frequencies (FOT) in term infants
Respiratory reactance (Xrs) - Term newborns | Postnatal day 3.
  Xrs at multiple frequencies (FOT) in term infants
Respiratory reactance (Xrs) - Term newborns | On the day of discharge
  Xrs at multiple frequencies (FOT) in term infants
Respiratory resistance (Rrs) - Preterm newborns | At NICU admission (within the first 2 hours).
  Rrs at multiple frequencies (FOT) in preterm infants
Respiratory resistance (Rrs) - Preterm newborns | Postnatal day 1.
  Rrs at multiple frequencies (FOT) in preterm infants
Respiratory resistance (Rrs) - Preterm newborns | Postnatal day 2.
  Rrs at multiple frequencies (FOT) in preterm infants
Respiratory resistance (Rrs) - Preterm newborns | Postnatal day 3.
  Rrs at multiple frequencies (FOT) in preterm infants
Respiratory resistance (Rrs) - Preterm newborns | On the first day of each additional week until 36 weeks post-conceptional age.
  Rrs at multiple frequencies (FOT) in preterm infants
Respiratory resistance (Rrs) - Preterm newborns | On the day of discharge.
  Rrs at multiple frequencies (FOT) in preterm infants
Respiratory reactance (Xrs) - Preterm newborns | At NICU admission (within the first 2 hours).
  Xrs at multiple frequencies (FOT) in preterm infants
Respiratory reactance (Xrs) - Preterm newborns | On postnatal day 1.
  Xrs at multiple frequencies (FOT) in preterm infants
Respiratory reactance (Xrs) - Preterm newborns | On postnatal day 2.
  Xrs at multiple frequencies (FOT) in preterm infants
Respiratory reactance (Xrs) - Preterm newborns | On postnatal day 3.
  Xrs at multiple frequencies (FOT) in preterm infants
Respiratory reactance (Xrs) - Preterm newborns | On the first day of each additional week until 36 weeks post-conceptional age.
  Xrs at multiple frequencies (FOT) in preterm infants
Respiratory reactance (Xrs) - Preterm newborns | On the day of discharge.
  Xrs at multiple frequencies (FOT) in preterm infants
Respiratory resistance (Rrs) - Infancy | At the age of 3 months (+/- 1 week)
  Rrs at multiple frequencies (FOT) during infancy
Respiratory resistance (Rrs) - Infancy | At the age of 6 months (+/- 1 week)
  Rrs at multiple frequencies (FOT) during infancy
Respiratory resistance (Rrs) - Infancy | At the age of 12 months (+/- 2 weeks)
  Rrs at multiple frequencies (FOT) during infancy
Respiratory reactance (Xrs) - Infancy | At the age of 3 months (+/- 1 week)
  Xrs at multiple frequencies (FOT) during infancy
Respiratory reactance (Xrs) - Infancy | At the age of 6 months (+/- 1 week)
  Xrs at multiple frequencies (FOT) during infancy
Respiratory reactance (Xrs) - Infancy | At the age of 12 months (+/- 2 weeks)
  Xrs at multiple frequencies (FOT) during infancy

CONTACTS AND LOCATIONS:
Overall Officials: Sotirios Fouzas, Principal Investigator — University of Patras
Locations (2):
- Greece (2):
  - Neonatal Intensive Care Unit, University Hospital of Patras, Pátrai
  - Well-baby nursery, Department of Pediatrics, University Hospital of Patras, Pátrai

IPD SHARING:
Plan to Share IPD: No
No Ethics Committee approval

REFERENCES:
- [Background] Skylogianni E, Douros K, Anthracopoulos MB, Fouzas S. The Forced Oscillation Technique in Paediatric Respiratory Practice. Paediatr Respir Rev. 2016 Mar;18:46-51. doi: 10.1016/j.prrv.2015.11.001. Epub 2015 Nov 10. PMID 26777151
- [Background] Hantos Z, Czovek D, Gyurkovits Z, Szabo H, Maar BA, Radics B, Virag K, Makan G, Orvos H, Gingl Z, Sly PD. Assessment of respiratory mechanics with forced oscillations in healthy newborns. Pediatr Pulmonol. 2015 Apr;50(4):344-52. doi: 10.1002/ppul.23103. Epub 2014 Aug 25. PMID 25154334
- [Background] Gray DM, Czovek D, McMillan L, Turkovic L, Stadler JAM, Vanker A, Radics BL, Gingl Z, Hall GL, Sly PD, Zar HJ, Hantos Z. Intra-breath measures of respiratory mechanics in healthy African infants detect risk of respiratory illness in early life. Eur Respir J. 2019 Jan 31;53(2):1800998. doi: 10.1183/13993003.00998-2018. Print 2019 Feb. PMID 30464010
- [Background] Klinger AP, Travers CP, Martin A, Kuo HC, Alishlash AS, Harris WT, Carlo WA, Ambalavanan N. Non-invasive forced oscillometry to quantify respiratory mechanics in term neonates. Pediatr Res. 2020 Aug;88(2):293-299. doi: 10.1038/s41390-020-0751-7. Epub 2020 Jan 14. PMID 31935746